CLINICAL TRIAL: NCT02806440
Title: Low Dose Naltrexone for Treatment of Pain in Patients With Fibromyalgia - Effect Via a Central Mechanism? A Randomized, Double-blinded, Placebo-controlled, Crossover Study.
Brief Title: Low Dose Naltrexone for Treatment of Pain in Patients With Fibromyalgia - Effect Via a Central Mechanism?
Acronym: LDN-in-FM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mads Werner, MD, PhD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-002972-26
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Low dose naltrexone; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose naltrexone (Active Comparator): Low dose naltrexone 4.5 mg/tablet, 1 tablet a day for 21 days
  Interventions: Drug: Low dose naltrexone
- Placebo (Placebo Comparator): Placebo tablet
  1 tablet a day for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose naltrexone — Active comparator
  Other Names: Naltrexone
  Arms: Low dose naltrexone
Drug: Placebo — Placebo comparator
  Other Names: Inert substance
  Arms: Placebo

SUMMARY:
This study evaluates the effect and mechanism of low dose naltrexone for treatment of pain in patients with fibromyalgia. It s a randomised, double-blinded, placebo-controlled, cross-over study.

The study takes place at The Multidisciplinary Pain Center in Grindsted.

DETAILED DESCRIPTION:
Fibromyalgia syndrome is a prevalent musculoskeletal disorder characterized by pain, profound fatigue, sleep disorder, mood disturbance etc. The prevalence is estimated to be 2-8%.

Treatment of pain in patients with fibromyalgia is often based on opioids. However, opioids may lead to tolerance, addiction and hyperalgesia and alternative treatments are therefore warranted.

Low dose naltrexone (3-5mg) (LDN) has shown promising results in the treatment of pain in patients with fibromyalgia, but there is a need for further research.

At the typical dose of naltrexone, 50 mg, it is an opioid antagonist. However LDN demonstrates analgesic and anti-inflammatory effects, possibly involving an antagonism of microglia in the CNS.

The investigators hypothesize, that LDN has a better pain relieving effect than placebo in in patients with fibromyalgia (FM). The investigators also hypothesize that LDN has a better effect upon experimentally induced pain in FM-patients, compared to placebo. A tentative mechanism is a central facilitation of the endogenous pain inbitory system.

ELIGIBILITY:
Patients diagnosed with fibromyalgia based on the criteria of American College of Rheumatology.

Inclusion Criteria:

* Widespread pain in patients with fibromyalgia (based on the above criteria)
* Enrolled as a patient in one of the multidisciplinary pain clinics involved in the project
* Inflammatory rheumatic disease (peripheral inflammation, including arthritis), must be excluded
* Women must be treated with a contraceptive measure, if not menopausal

Exclusion Criteria:

* Cancer
* Treatment with opioids (other analgesic treatments in stabile dose 14 days prior to study start are allowed)
* Change in stabile treatment (p.n. paracetamol is allowed, but must be registered)
* Pregnant/breastfeeding
* Does not speak/understand Danish
* Allergy to the ingredient
* Severe liver impairment
* Severe kidney impairment
* Acute hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in pain scores (during rest, during household activity, during personal daily hygienic procedures) | Baseline: Day -2 to day 1 (baseline before treatment 1); Treatment 1: Day 19 to 21 ; Washout: Day 33 to 35 (baseline before treatment 2); Treatment 2: Day 54 to 56
  The patient indicates using a questionnaire-based numerical rating scale (0 = no pain; 100 = worst imaginable pain) mean values of pain at rest, pain during household activity and pain during personal hygienic procedures in the preceding 24 hrs. The cumulated pain scores are used in the statistical analyses.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised (FIQR) | Before baseline: Day -3; Treatment 1: Baseline (Day 1) + Day 14 + 21 ; Washout: Before baseline day -3; Treatment 2: Baseline (Day 35) + Day 49 + 56
  The FIQR is a fibromyalgia-specific questionnaire containing three domains: function domain, impact domain and symptom domain. The total score of FIQR is calculated by:
  * the function domain sum is divided by 3 (upper limit 30)
  * the impact domain sum is unchanged (upper limit 20)
  * the symptom domain sum is divided by 2 (upper limit 50) The three resulting processed domain scores are summed to obtain the total score of the FIQR (range 0-100)
Daily Sleep Interference Scale (DSIS) | Diary (Treatment 1: baseline (Day 1) to Day 21; Treatment 2: baseline (Day 35) to Day 56)
  Pain-related sleep interference is evaluated with the DSIS (0 =pain does not interfere with sleep, 10 = pain completely interferes with sleep]).
Pressure algometry (1 sq.cm probe) | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  Pressure algometry in pre-specified points:
  1. right occipital region at insertion of m. subocipitalis
  2. right m. trapezius at the midpoint of the upper border
  3. right paraspinal region, 3 cm lateral of the midline at level of mid-scapula
  4. right second costochondral junction
  5. right lateral epicondyle
  6. right knee region, at the medial "fat pad" proximal of the meniscus margin
  In addition at following control sites:
  1. right lower arm, at the dorsal lower third
  2. right fingernail of first digit
  3. right third metatarsal bone at midpoint Cut-off point is 400 kPa, rate 10-30 kPa/s
Hospital Anxiety and Depression Scale (HADS) | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  HADS is a 14-item questionnaire used to evaluate the subject's level of anxiety and depression; the subjects can rate between 0-21 with a score of eleven as the cutoff point for anxiety or depression
Pain Catastrophizing Scale (PCS) | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  The PCS is a 13-item self-report scale to measure pain catastrophizing: each item is rated on a 5-point nominal scale (0 = not at all, 4 = all the time). It is constructed with three subscales being magnification, rumination, and helplessness.
Adverse effects | Diary + Treatment 1: Baseline (day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  Self-reported adverse effects related to the treatment:
  CNS: irritability, mood changes, drowsiness, lethargy, sleep dysfunction, dizziness cardiovascular system: palpitations, orthostatic hypotension g.i.-system: dyspepsia, nausea, obstipation, diarrhoea urogenital system: urinary retention, urinary incontinence autonomic system: diaphoresis, shivering
Quantitative Sensory Testing (QST) | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  Cold pressor test (1min, 10C) - Pressure tolerance threshold before and after Cold Water.
  Heat/Capsaicin test - 5min, 45C heat, followed by 30min capsaicin cream 0.075%, Measurement of allodynic (brush, Somedic) and hyperalgesic (Pinprick stimulator 128nm) areas.
Plasma concentrations of naltrexone and β-Naltrexon | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
Pain DETECT | Treatment 1: Baseline (Day 1) + Day 14 + Day 21; Treatment 2: Baseline (Day 35) + Day 49 + Day 56
  Measurement of neuropathic component
Brief Pain Inventory - Short Form (BPI-SF) questionnaire | Before baseline: Day -3 to -1; Washout: Before baseline Day 32 to 34
  BPI-SF allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function.
  BPI-SF is a widely used Measurement Tool for assessing clinical pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten M Bested, MD, Principal Investigator — Multidisciplinary Pain Clinic
Locations (1):
- Multidisciplinary Pain Centre, Grindsted, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be made available in a public research database as part of the final publication.

REFERENCES:
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Gilron I, Jensen TS, Dickenson AH. Combination pharmacotherapy for management of chronic pain: from bench to bedside. Lancet Neurol. 2013 Nov;12(11):1084-95. doi: 10.1016/S1474-4422(13)70193-5. Epub 2013 Sep 25. PMID 24074723
- [Background] Younger J, Parkitny L, McLain D. The use of low-dose naltrexone (LDN) as a novel anti-inflammatory treatment for chronic pain. Clin Rheumatol. 2014 Apr;33(4):451-9. doi: 10.1007/s10067-014-2517-2. Epub 2014 Feb 15. PMID 24526250
- [Result] Younger JW, Zautra AJ, Cummins ET. Effects of naltrexone on pain sensitivity and mood in fibromyalgia: no evidence for endogenous opioid pathophysiology. PLoS One. 2009;4(4):e5180. doi: 10.1371/journal.pone.0005180. Epub 2009 Apr 13. PMID 19365548
- [Result] Younger J, Noor N, McCue R, Mackey S. Low-dose naltrexone for the treatment of fibromyalgia: findings of a small, randomized, double-blind, placebo-controlled, counterbalanced, crossover trial assessing daily pain levels. Arthritis Rheum. 2013 Feb;65(2):529-38. doi: 10.1002/art.37734. PMID 23359310